CLINICAL TRIAL: NCT03719144
Title: Optimizing Anticoagulation Dosing and Adherence for Patients With Non-valvular Atrial Fibrillation
Brief Title: Understanding and Improving Anticoagulation Dosing for Patients With Atrial Fibrillation
Acronym: ARISTA
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00088597
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients registered on ResearchMatch.org with Atrial Fibrillation as a medical condition; or who participate in afib-related social media platforms and confirm a diagnosis of afib, will be invited to participate in this study. Patients will be consented using an online consent form and then will be asked to complete 1 survey that contains scenarios and ranking questions.
- Providers: Providers who have contributed at least 25 Atrial Fibrillation patients to the Symphony pharmacy claims dataset will be contacted to participate. Interested providers will be consented using an online consent form and then will be asked to complete 1 survey that contains scenarios and ranking questions.

SUMMARY:
This study will survey atrial fibrillation patients to better understand patient perspective of DOAC treatment, and providers to assess knowledge, practice patterns, and beliefs surrounding anticoagulation for AF.

ELIGIBILITY:
Inclusion Criteria:

Retrospective Analysis:

1. NVAF documented in at least 2 claims between January 2015 and December 2016
2. CHA2DS2-VASc scores of 2 or higher

Prospective Analysis:

1. Patient Analysis: All patients in ResearchMatch with diagnosed AF.
2. Provider Analysis: All providers who contributed at least 25 AF patients treated with DOACs to the Symphony claims dataset. All provider specialties (i.e. cardiology, primary care, and other), as well as provider types (i.e. physician, physician extender, and nurse practitioner) will be included.

Exclusion Criteria:

Retrospective Analysis:

1. Patients with bioprosthetic or mechanical valves in the mitral position.
2. Patients with any of the following missing data: age, sex, body weight, serum creatinine, and any data required for DOAC dosing.
3. Patients with mitral stenosis.
4. Patients without 12-month follow-up data.

Prospective Analysis:

1. Provider Analysis: All providers who contributed less than 25 AF patients treated with DOACs to the Symphony claims dataset.
2. Patient Analysis: Patients unwilling or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is targeting AF patients and providers.
Sampling Method: Non-Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
The co-primary outcome for the retrospective analysis is rate of 12-month medication discontinuation. | up to 12 months
  The pharmacy claims dataset will be used to obtain records of patient prescription fills, and the characteristics of those patients filling the prescriptions. The index event for each patient will be defined by when the second NVAF claim was filed. The dose will be initially determined from the index prescription. Of those patients prescribed a DOAC, the 12-month DOAC discontinuation rates will be examined. DOAC discontinuation will be defined as a gap in fill ≥30 days following the run-out date of the last observed claim for the index therapy. Twelve-month DOAC discontinuation will be stratified according to whether the patient received a dose reduction following labeled criteria, a dose reduction inconsistent with labeled criteria, or were prescribed the full dose, per labeled criteria.
The co-primary outcome for the retrospective analysis is 12-month adherence rates. | up to 12 months
  The pharmacy claims dataset will be used to obtain records of patient prescription fills, and the characteristics of those patients filling the prescriptions. The index event for each patient will be defined by when the second NVAF claim was filed. The dose will be initially determined from the index prescription. Of those patients prescribed a DOAC, medication adherence rates will be examined. DOAC adherence, defined as the proportion of days covered ≥80%, is calculated by the number of days any anticoagulant is available divided by the number of days in the follow-up period. Twelve-month adherence rates will be stratified according to whether the patient received a dose reduction following labeled criteria, a dose reduction inconsistent with labeled criteria, or were prescribed the full dose, per labeled criteria.

OTHER OUTCOMES:
Prevalence of under-dosing | up to 12 months
  Providers who contributed at least 25 NVAF patients on DOACs to the pharmacy claims dataset will be grouped into tertiles based on the frequency of under-dosing: high, intermediate, and low. We will examine the association of provider factors with the likelihood of under-dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Y Wang, MD, Principal Investigator — Duke Clinical Research Institute, Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Analysis of Oral Anticoagulant Dosing and Adherence to Therapy Among Patients With Nonvalvular Atrial Fibrillation — https://pubmed.ncbi.nlm.nih.gov/37285155/
- See also: Differences in Preferences Between Clinicians and Patients for the Use and Dosing of Direct Oral Anticoagulants for Atrial Fibrillation — https://pubmed.ncbi.nlm.nih.gov/33998252/